CLINICAL TRIAL: NCT03141333
Title: A Randomized Feasibility Trial Evaluating a Teleintervention for Families of Children With Developmental Coordination Disorder (DCD)
Brief Title: A Teleintervention in Developmental Coordination Disorder
Acronym: DCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: usherbrooke
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-01

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleintervention (Experimental): Participants of this group will have access to the following sections in the web plate-form: information, forum, chat and live online consultation. The teleintervention consists of having access to the forum, chat and live online consultation sections of the web plate-form.
  Interventions: Behavioral: Teleintervention
- No intervention (No Intervention): Participants of this group will have access to the following section of the web plate-form: information, which is consistent with the standard of care for many families of children with DCD, who only have access to online information but do not have access to any type of intervention.

INTERVENTIONS:
Behavioral: Teleintervention — Participants of this group will have access to the following sections in the web plate-form: information, forum, chat and live online consultation. The teleintervention consists of having access to the forum, chat and live online consultation sections of the web plate-form.
  Arms: Teleintervention

SUMMARY:
The principal study goals are to determine if a randomized control trial would be feasible, particularly with regards to i) recruitment and retention of parents of children having a diagnosis or a suspicion of diagnosis of DCD, and ii) parents' utilization of the teleintervention. The study will also examine quantitatively and qualitatively families' acceptability of- and satisfaction with the teleintervention.

DETAILED DESCRIPTION:
Developmental coordination disorder (DCD) is a neurodevelopmental disorder characterised by difficulties in planning and execution of motor coordination activities like dressing, sports and writing. Increasing parents' capacity to manage their children's needs is part of the recommended DCD best practices, as soon as children are suspected to have DCD or early following diagnosis. Parents' capacity could be increased through simple, community-based interventions using a consultative approach. Using the Internet could be an interesting avenue to develop public community-based services and build parents' capacity to manage their child with DCD. The feasibility of recruiting and using the Internet to build parents' capacity is however unknown, since no such study have been conducted.

This randomized feasibility trail will experiment a teleintervention, characterized by a virtual interaction between a health professional and a user by Internet, for children with DCD. The principal study goals are to determine if a randomized control trial would be feasible, particularly with regards to i) recruitment and retention of parents of children having a diagnosis or a suspicion of diagnosis of DCD, and ii) parents' utilization of the teleintervention. The study will also examine quantitatively and qualitatively families' acceptability of- and satisfaction with the teleintervention. As part of the evaluation of acceptability, the impact of the teleintervention on parental competencies will be explored. At the end of the 3-months randomized feasibility trial, the influence of the number of participants on the utilization of the teleintervention will be explored by providing access to the teleintervention to all participants (control and intervention).

ELIGIBILITY:
Inclusion Criteria:

* A DCD medical diagnostic (or DCD medical hypothesis)
* Must be at or under the 16e percentile for the global score at the Movement Assessment Battery for Children-2 (MABC-2) or be at or under the 5e for one of the 3 subscale of the MABC-2.

Exclusion Criteria:

* Do not have other neurodevelopmental diagnoses, with the exception of Attention Deficit Hyperactivity Disorder (ADHD)
* Do not receive rehabilitation services for DCD in the public health care system

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Utilization of the teleintervention | 3 months (from day 1 to study completion)
  Time spent on the web plate-form (calculated in minutes, time spent on the plate-form during the 3 months teleintervention)

SECONDARY OUTCOMES:
Recruitment and retention | Number of participants at baseline and at completion of the study (3 months later)
  Number of participants recruited and retention rate
Parents' sense of competencies | Collected at baseline and at completion of the study (3 months later)
  Parenting Sense of Competence Scale
Parents' satisfaction with the intervention | At completion of the study (3 months following the begining of the teleintervention)
  Qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Camden, Principal Investigator — CR CHUS
Locations (1):
- CR CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No